CLINICAL TRIAL: NCT04193904
Title: A Safety and Preliminary Efficacy Study of the Oral Live Biotherapeutic MRx0518 With Hypofractionated Preoperative Radiation for Resectable Pancreatic Cancer
Brief Title: A Study of Live Biotherapeutic Product MRx0518 With Hypofractionated Radiation Therapy in Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor insolvency
Sponsor: 4D pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRx0518-I-003
Record Dates: First submitted 2019-11-12; First posted 2019-12-10 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRx0518 with hypofractionated preoperative radiation (Experimental): Subjects will take one capsule of MRx0518 twice daily from one week prior to radiation therapy until surgical resection (6 to 9 weeks approx.) Radiation therapy will be delivered as 30Gy/10 fractions over 2 weeks.
  Interventions: Drug: MRx0518; Radiation: Hypofractionated Preoperative Radiation

INTERVENTIONS:
Drug: MRx0518 — MRx0518 is a live biotherapeutic product consisting of a lyophilised formulation of a proprietary strain of bacterium. The study dosing regimen is one capsule two times per day for the duration of the treatment period.
Radiation: Hypofractionated Preoperative Radiation — Radiation will be delivered as 30Gy/10 fractions over two weeks.

SUMMARY:
This is a single center, open-label, phase I study to evaluate the safety and preliminary efficacy of MRx0518 with preoperative hypofractionated radiation in 15 patients with resectable pancreatic cancer.

Subjects will take MRx0518 daily for one week prior to the start of radiation therapy, throughout radiation and until surgical resection of the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed informed consent and is willing to comply with the protocol
* Cytologic or biopsy confirmed adenocarcinoma of the pancreas
* TNM stage: Tx, T1-4, N0-1 or Nx, M0
* Potentially resectable pancreatic cancer defined as no extra-pancreatic disease, no evidence of tumor extension to the celiac axis, common hepatic artery and superior mesenteric artery, and no evidence of deformity of the superior mesenteric vein or superior mesenteric portal vein confluence
* No evidence of distant metastases either prior to or after induction chemotherapy
* Able to comply with instructions required for radiation therapy
* Age 18 years or older
* Completion of 2-6 months of standard induction chemotherapy (mFOLFIRINOX, gemcitabine and nab-paclitaxel or other)
* Eastern Cooperative Oncology Group Score 0, 1 or 2
* Adequate haematologic function (absolute neutrophil count ≥1500mm3; haemoglobin ≥8.0 g/dL; platelet count ≥50000mm3)
* Adequate renal and liver function (creatinine ≤ 1.5 x upper limit of normal; total bilirubin ≤ 1.5 x upper limit of normal; aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal; alkaline phosphatase ≤ 2.5 x upper limit of normal

Exclusion Criteria:

* Prior radiation therapy to the abdomen that would overlap with the treatment field
* Prior surgical resection of pancreatic tumor
* Receiving any approved or investigational anti-cancer agent other than those provided for in this study
* Uncontrolled or active gastric or duodenal ulcer disease within 30 days of dosing
* Residual or ongoing ≥Grade 3 toxicity from chemotherapy
* Contraindication to IV contrast that can't be managed with pre-medication
* Concurrent participation in another interventional clinical trial or use of another investigational agent within 30 days of consent (concurrent non-interventional trials are eligible)
* Uncontrolled intercurrent illness including but not limited to, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia, stroke, or psychiatric illness that would limit compliance with treatment
* Second primary malignancy within the last 5 years, unless treated definitively and/or low risk in the judgement of the treating investigator
* Known history of HIV or active hepatitis B/C (patients who have been vaccinated for hepatitis B and do not have history of infection are eligible)
* Known intolerance or hypersensitivity to study drug
* Subjects who are allergic to amoxicillin/clavulanic acid, erythromycin and imipenem
* Female subjects who are breastfeeding
* Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control for the entire study and for 30 days after last dose of MRx0518. A negative pregnancy test must be obtained within 14 days prior to start of treatment
* Male subjects who are unwilling or unable to use an acceptable method of birth control for the entire study period and for 30 days after last dose of MRx0518
* Serious infection requiring systemic therapy
* Use of systemic antibiotics within 2 weeks of start of study treatment
* Has a known inability for intake of oral capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety of MRx0518 in combination with hypofractionated preoperative radiation through the collection of adverse events | Up to 1 year post completion of radiation
  Adverse events will be assessed as per CTCAE v5.0

SECONDARY OUTCOMES:
Major pathologic response | At time of surgery
  Major pathologic response is defined as <5% viable cells in resected tumour specimen
Tumour infiltrating lymphocytes (TILs) | Baseline to Surgery
  Changes in TILs from optional baseline biopsy to resected tumour specimen will be assessed.
Overall Survival (OS) | 12 months post radiation
  OS is defined as the duration from the start of study treatment until death due to any cause
Progression Free Survival (PFS) | 12 months post radiation
  PFS is defined as the duration from the start of study treatment until disease progression or death
Local Control | 6 months post radiation
  Local control is defined as absence of progression at the primary site and will be assessed with imaging
Distant Control | 6 months post radiation
  Distant control is defined as absence of progression at any site other than the primary site and will be assessed with imaging
Margin status | At time of surgery
  The margin status of the tumour at the time of surgery will be assessed

OTHER OUTCOMES:
Changes to microbiome | Baseline to 6 months post completion of radiation
  The microbiome profile of faecal, urine, tumour and duodenum samples will be analysed for changes using the MicroDx platform
Tumour immune infiltration | Baseline to Surgery
  Optional biopsies and resection specimens will be assessed for changes in tumour immune infiltrates
Landscape of immune and stromal cells | Baseline to Surgery
  Optional biopsy and resection specimens will be catalogued for the landscape of immune and stromal cells
Changes in Circulating Tumour Cells | Baseline to 6 months post completion of radiation
  Blood samples will be assessed for presence of circulating tumour cells, circulating tumour DNA and/or circulating immune cells
Genomic changes | Baseline to 6 months post completion of radiation
  Whole exome sequencing and transcriptome sequencing from tumour and blood samples will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Cullen M Taniguchi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No